CLINICAL TRIAL: NCT04293705
Title: Congenital Disability and Rehabilitation of Cognitive and Behavioral Difficulties by Using the Teen Online Problem-Solving (TOPS) Program.
Brief Title: Congenital Disability and Rehabilitation: the TOPS Program
Acronym: TOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 350
Record Dates: First submitted 2020-02-25; First posted 2020-03-03 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2021-06

CONDITIONS: Congenital Disorders
Keywords: Congenital Disorders
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Intervention Model Description: Group 1 performs the regular TOPS intervention on problem-solving and executive function-related behaviors, while Group 2, serving as active control group, performs a modified version of the TOPS including only sessions on health and wellness but no contents on problem-solving and executive function-related behaviors.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Outcomes assessors and participants are blinded with respect to group assignment, as both Group 1 and Group 2 use the TOPS program platform, even though with different contents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- regular TOPS group (Experimental): Patients are required to perform the regular TOPS program, composed of 10 core sessions and other eventual supplementary sessions. In addition, biweekly Google Meet sessions with a cognitive-behavioral psychotherapist are scheduled, with the aim to monitor patients' activities on problem-solving related to the TOPS program contents and the problem solving process in real life. The program has a specific focus on problem-solving, executive functions, behavioral strategies and social skills.
  Interventions: Device: Teen On-line Problem Solving
- modified TOPS group (Active Comparator): Patients are required to perform the modified TOPS program, composed of 10 sessions focused only on health and wellness contents. Thus, this program does not include contents on problem-solving, executive functions, behavioral strategies and social skills, representing a low cognitively simulating activity. Biweekly Google Meet sessions with a cognitive-behavioral psychotherapist are scheduled, with the aim of monitoring training adherence and discuss the program's contents.
  Interventions: Device: Teen On-line Problem Solving

INTERVENTIONS:
Device: Teen On-line Problem Solving — The TOPS program is a web-based platform delivered on computers and tablets, which is composed of different self-guided, online sessions on different contents: executive functions, social skills, behavioral strategies, injury-related issues and health and wellness. The TOPS program has been designed to be performed by patients and their families at home. Biweekly Google Meet videoconferences between a coach with expertise in cognitive-behavioral psychotherapy and patients are scheduled along the entire duration of the program.
  Other Names: TOPS

SUMMARY:
The study aims at evaluating the feasibility and the efficacy of the Teen On-line Problem Solving program (TOPS) in improving executive functioning and behavior problems in adolescents aged 11-19 years with congenital disability due to brain malformation/syndrome.

In order to control for placebo effects, participants are randomized into two intervention conditions. Group 1 performs the regular version of the TOPS, while Group 2 performs a modified version containing no activities on executive functions, behavioral strategies and social skills.

DETAILED DESCRIPTION:
Adolescents with congenital brain malformation/syndrome often present with executive dysfunction and behavioral and social problems. Ad hoc rehabilitation may significantly ameliorate such difficulties. With this aim, the Teen On-line Problem-Solving program (TOPS) could represent a suitable opportunity of intervention, as it aims at helping children to improve executive and behavioral functioning. The program consists of a web-based platform composed of 10 core sessions and eventual supplementary sessions, providing information and activities on executive functioning, behavioral strategies, social skills and injury-related issues and health and wellness. The program is delivered remotely, with patients performing the intervention at home, together with their families. Biweekly Google Meet sessions with a cognitive-behavioral psychotherapist are scheduled along the entire duration of the intervention to monitor the activities related to the program and the real-life problem-solving process that patients are required to perform during the intervention.

Assessment of executive functions and behavioral problems is conducted before and after the training (immediate post training assessment and follow-up assessment 6 months after the end of the training), in order to investigate the presence of significant changes after the intervention. Both questionnaires and performance-based measures are used.

Participants are randomized into two groups: Group 1 performs the regular version of the TOPS, while Group 2 performs a modified version containing no activities on executive functions, behavioral strategies and social skills.

Based on the average effect of TOPS program reported by a meta-analysis available in the literature (Corti et al., 2019; Hedge's g = 0.39) we estimated a small-to-moderate effect size of f =0.2 (f was calculated based on Hedge's g value). Power analysis was conducted by using GPower3 software. Assuming a correlation of 0.50 between repeated measures and setting the alfa level at P < 0.05, a sample size of 21 subjects per group is required to obtain 80% of power with our 2 groups x 3 time points design.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of congenital disability due to brain malformation/syndrome

Exclusion Criteria:

* history of abuse
* familiarity for psychiatric hospitalization

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Behavior Rating Inventory of Executive Function Second Edition (BRIEF 2) - parent form - baseline | baseline (immediately pre-training)
  The BRIEF questionnaire is aimed at assessing executive functioning at home and school and contains 63 items in different clinical scales and validity scales. The questionnaire is administered to parents, which have to rate the frequency of dysexecutive problems of their children on a 3-point Likert Scale. Raw scores of the global scale range from 63 to 189. T scores (M = 50, SD = 10) are used to interpret the level of executive functioning. Higher scores mean a worse outcome.
Behavior Rating Inventory of Executive Function Second Edition (BRIEF 2) - parent form - change at 6 months (immediately post-training) | post-training (approximatively at month 6)
  The BRIEF questionnaire is aimed at assessing executive functioning at home and school and contains 63 items in different clinical scales and validity scales. The questionnaire is administered to parents, which have to rate the frequency of dysexecutive problems of their children on a 3-point Likert Scale. Raw scores of the global scale range from 63 to 189. T scores (M = 50, SD = 10) are used to interpret the level of executive functioning. Higher scores mean a worse outcome.
Behavior Rating Inventory of Executive Function Second Edition (BRIEF 2) - parent form - change at 12 months (follow-up at 6 months after the end of the training) | follow-up (approximatively at month 12)
  The BRIEF questionnaire is aimed at assessing executive functioning at home and school and contains 63 items in different clinical scales and validity scales. The questionnaire is administered to parents, which have to rate the frequency of dysexecutive problems of their children on a 3-point Likert Scale. Raw scores of the global scale range from 63 to 189. T scores (M = 50, SD = 10) are used to interpret the level of executive functioning. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Function Second Edition (BRIEF 2) - self report form - baseline | baseline (immediately pre-training)
  The BRIEF questionnaire is aimed at assessing self-reported executive functioning at home and school of adolescents aged 11-18 years and contains 55 items in different clinical scales and validity scales. Raw scores of the global scale range from 55 to 165. T scores (M = 50, SD = 10) are used to interpret the level of executive functioning. Higher scores mean a worse outcome.
Behavior Rating Inventory of Executive Function Second Edition (BRIEF 2) - self report form - change at 6 months | post-training (approximatively at month 6)
  The BRIEF questionnaire is aimed at assessing self-reported executive functioning at home and school of adolescents aged 11-18 years and contains 55 items in different clinical scales and validity scales. Raw scores of the global scale range from 55 to 165. T scores (M = 50, SD = 10) are used to interpret the level of executive functioning. Higher scores mean a worse outcome.
Behavior Rating Inventory of Executive Function Second Edition (BRIEF 2) - self report form - change at 12 months | post-training (approximatively at month 12)
  The BRIEF questionnaire is aimed at assessing self-reported executive functioning at home and school of adolescents aged 11-18 years and contains 55 items in different clinical scales and validity scales. Raw scores of the global scale range from 55 to 165. T scores (M = 50, SD = 10) are used to interpret the level of executive functioning. Higher scores mean a worse outcome.
Child Behavior Checklist 6-18 (CBCL 6-18) - baseline | baseline (immediately pre-training)
  The CBCL 6-18 is aimed at assessing psychological adjustment and behavioral functioning of children, as rated by parents. This instrument provides a total score, an internalizing score and an externalizing score, together with 8 syndrome scale scores and 6 DSM-oriented scale scores. It contains 113 items. Raw scores of the Total Problems Scale range from 0 to 226. T scores (M = 50, SD = 10) are used to interpret the level of behavioral functioning. Higher scores mean a worse outcome.
Child Behavior Checklist 6-18 (CBCL 6-18) - change at 6 months | post-training (approximatively at month 6)
  The CBCL 6-18 is aimed at assessing psychological adjustment and behavioral functioning of children, as rated by parents. This instrument provides a total score, an internalizing score and an externalizing score, together with 8 syndrome scale scores and 6 DSM-oriented scale scores. It contains 113 items. Raw scores of the Total Problems Scale range from 0 to 226. T scores (M = 50, SD = 10) are used to interpret the level of behavioral functioning. Higher scores mean a worse outcome.
Child Behavior Checklist 6-18 (CBCL 6-18) - change at 12 months | post-training (approximatively at month 12)
  The CBCL 6-18 is aimed at assessing psychological adjustment and behavioral functioning of children, as rated by parents. This instrument provides a total score, an internalizing score and an externalizing score, together with 8 syndrome scale scores and 6 DSM-oriented scale scores. It contains 113 items. Raw scores of the Total Problems Scale range from 0 to 226. T scores (M = 50, SD = 10) are used to interpret the level of behavioral functioning. Higher scores mean a worse outcome.
Youth Self-Report 11-18 (YSR 11-18) - baseline | baseline (immediately pre-training)
  YSR 11-18 is aimed at assessing self-reported psychological adjustment and behavioral functioning of adolescents aged 11-18 years. This instrument provides a total score, an internalizing score and an externalizing score, together with eight empirically based syndromes and DSM-oriented scales. It contains 112 items. Raw scores of the Total Problems Scale range from 0 to 224. T scores (M = 50, SD = 10) are used to interpret the level of behavioral functioning. Higher scores mean a worse outcome.
Youth Self-Report 11-18 (YSR 11-18) - change at 6 months | post-training (approximatively at month 6)
  YSR 11-18 is aimed at assessing self-reported psychological adjustment and behavioral functioning of adolescents aged 11-18 years. This instrument provides a total score, an internalizing score and an externalizing score, together with eight empirically based syndromes and DSM-oriented scales. It contains 112 items. Raw scores of the Total Problems Scale range from 0 to 224. T scores (M = 50, SD = 10) are used to interpret the level of behavioral functioning. Higher scores mean a worse outcome.
Youth Self-Report 11-18 (YSR 11-18) - change at 12 months | post-training (approximatively at month 12)
  YSR 11-18 is aimed at assessing self-reported psychological adjustment and behavioral functioning of adolescents aged 11-18 years. This instrument provides a total score, an internalizing score and an externalizing score, together with eight empirically based syndromes and DSM-oriented scales. It contains 112 items. Raw scores of the Total Problems Scale range from 0 to 224. T scores (M = 50, SD = 10) are used to interpret the level of behavioral functioning. Higher scores mean a worse outcome.
Back Anxiety Inventory (BAI) - baseline | baseline (immediately pre-training)
  BAI is a 21-item questionnaire aimed at assessing state and trait anxiety. In this study the questionnaire is administered to parents to evaluate their psychological functioning. The total score is calculated by finding the sum of the 21 items (4-point Likert scale ranging from 0 to 3), with a minimum score of 0 and a maximum score of 108. Higher scores mean a worse outcome. Score of 0-21 indicates low anxiety; score of 22-35 indicates moderate anxiety; score of 36 and above (maximum: 108) indicates potentially concerning levels of anxiety.
Back Anxiety Inventory (BAI) - change at 6 months | post-training (approximatively at month 6)
  BAI is a 21-item questionnaire aimed at assessing state and trait anxiety. In this study the questionnaire is administered to parents to evaluate their psychological functioning. The total score is calculated by finding the sum of the 21 items (4-point Likert scale ranging from 0 to 3), with a minimum score of 0 and a maximum score of 108. Higher scores mean a worse outcome. Score of 0-21 indicates low anxiety; score of 22-35 indicates moderate anxiety; score of 36 and above (maximum: 108) indicates potentially concerning levels of anxiety.
Back Anxiety Inventory (BAI) - change at 12 months | post-training (approximatively at month 12)
  BAI is a 21-item questionnaire aimed at assessing state and trait anxiety. In this study the questionnaire is administered to parents to evaluate their psychological functioning. The total score is calculated by finding the sum of the 21 items (4-point Likert scale ranging from 0 to 3), with a minimum score of 0 and a maximum score of 108. Higher scores mean a worse outcome. Score of 0-21 indicates low anxiety; score of 22-35 indicates moderate anxiety; score of 36 and above (maximum: 108) indicates potentially concerning levels of anxiety.
Symptom Checklist 90 (SCL-90) - baseline | baseline (immediately pre-training)
  The SCL-90 is a self-report questionnaire aimed at measuring psychiatric symptom intensity on nine different subscales. The 90 items are scored on a five-point Likert scale (ranging from 0 to 4), indicating the rate of occurrence of the symptoms during the last 7 days. In this study the questionnaire is administered to parents to assess parental psychological distress, by considering the Global Severity Index (GSI). Raw scores of the GSI, which are calculated as the average score of the 90 items of the questionnaire, range from 0 to 360. The final score is reported as T score (M = 50 SD = 10). Higher scores indicate higher distress. Consistent with the recommendations of Derogatis (1994), a T score at or above 63 on the GSI indicates the clinical range.
Symptom Checklist 90 (SCL-90) - change at 6 months | post-training (approximatively at month 6)
  The SCL-90 is a self-report questionnaire aimed at measuring psychiatric symptom intensity on nine different subscales. The 90 items are scored on a five-point Likert scale (ranging from 0 to 4), indicating the rate of occurrence of the symptoms during the last 7 days. In this study the questionnaire is administered to parents to assess parental psychological distress, by considering the Global Severity Index (GSI). Raw scores of the GSI, which are calculated as the average score of the 90 items of the questionnaire, range from 0 to 360. The final score is reported as T score (M = 50 SD = 10). Higher scores indicate higher distress. Consistent with the recommendations of Derogatis (1994), a T score at or above 63 on the GSI indicates the clinical range.
Symptom Checklist 90 (SCL-90) - change at 12 months | post-training (approximatively at month 12)
  The SCL-90 is a self-report questionnaire aimed at measuring psychiatric symptom intensity on nine different subscales. The 90 items are scored on a five-point Likert scale (ranging from 0 to 4), indicating the rate of occurrence of the symptoms during the last 7 days. In this study the questionnaire is administered to parents to assess parental psychological distress, by considering the Global Severity Index (GSI). Raw scores of the GSI, which are calculated as the average score of the 90 items of the questionnaire, range from 0 to 360. The final score is reported as T score (M = 50 SD = 10). Higher scores indicate higher distress. Consistent with the recommendations of Derogatis (1994), a T score at or above 63 on the GSI indicates the clinical range.
Parenting Stress Index (PSI) - Short Form - baseline | baseline (immediately pre-training)
  PSI - Short Form is a 36-item questionnaire aimed at assessing levels of stress associated with parenting. The 36 items are scored on a five-point Likert scale. PSI - Short Form is directly administered to parents. A global score (PSI-total) and three subscales, namely Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI) and Difficult Child (DC), are provided. The clinical cut-off of PSI-total is established at 90 (Abidin 2008). Higher scores indicate higher distress.
Parenting Stress Index (PSI) - Short Form - change at 6 months | post-training (approximatively at month 6)
  PSI - Short Form is a 36-item questionnaire aimed at assessing levels of stress associated with parenting. The 36 items are scored on a five-point Likert scale. PSI - Short Form is directly administered to parents. A global score (PSI-total) and three subscales, namely Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI) and Difficult Child (DC), are provided. The clinical cut-off of PSI-total is established at 90 (Abidin 2008). Higher scores indicate higher distress.
Parenting Stress Index (PSI) - Short Form - change at 12 months | post-training (approximatively at month 12)
  PSI - Short Form is a 36-item questionnaire aimed at assessing levels of stress associated with parenting. The 36 items are scored on a five-point Likert scale. PSI - Short Form is directly administered to parents. A global score (PSI-total) and three subscales, namely Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI) and Difficult Child (DC), are provided. The clinical cut-off of PSI-total is established at 90 (Abidin 2008). Higher scores indicate higher distress.
Jansari Assessment of Executive Functioning - Adolescents (JEF-A) - baseline | baseline (immediately pre-training)
  JEF-A is an ecologically-valid computerized assessment using non-immersive virtual reality aimed at evaluating executive functions in adolescents. It is a performance-based assessment. Participants are asked to plan, set up and run a birthday party through the completion of 16 tasks resembling real-world activities. All tasks are scored on a 3-point scale: 0 for failure, 1 for a partial or nonoptimal completion, and 2 for satisfactory completion. The final raw score ranges from 0 to 32. Higher scores mean a better executive functioning.
Jansari Assessment of Executive Functioning - Adolescents (JEF-A) - change at 6 months | post-training (approximatively at month 6)
  JEF-A is an ecologically-valid computerized assessment using non-immersive virtual reality aimed at evaluating executive functions in adolescents. It is a performance-based assessment. Participants are asked to plan, set up and run a birthday party through the completion of 16 tasks resembling real-world activities. All tasks are scored on a 3-point scale: 0 for failure, 1 for a partial or nonoptimal completion, and 2 for satisfactory completion. The final raw score ranges from 0 to 32. Higher scores mean a better executive functioning.
Jansari Assessment of Executive Functioning - Adolescents (JEF-A) - change at 12 months | post-training (approximatively at month 12)
  JEF-A is an ecologically-valid computerized assessment using non-immersive virtual reality aimed at evaluating executive functions in adolescents. It is a performance-based assessment. Participants are asked to plan, set up and run a birthday party through the completion of 16 tasks resembling real-world activities. All tasks are scored on a 3-point scale: 0 for failure, 1 for a partial or nonoptimal completion, and 2 for satisfactory completion. The final raw score ranges from 0 to 32. Higher scores mean a better executive functioning.
A Developmental NEuroPSYchological Assessment-II (NEPSY-II) (Theory of Mind and Emotion Recognition subscales) - baseline | baseline (immediately pre-training)
  The Theory of Mind and Affect Recognition subscales of NEPSY II are performance-based subtests aimed at evaluating social perception. They are administered to adolescents. Theory of Mind subscale-part A raw scores range from 0 to 17, Theory of Mind subscale-part b raw scores range from 0 to 8. Theory of Mind total subscale raw scores range from 0 to 25. Affect Recognition subscale raw scores range from 0 to 35. Raw scores are converted in scaled scores ranging from 1 to 19. Higher scores mean better outcomes.
A Developmental NEuroPSYchological Assessment-II (NEPSY-II) (Theory of Mind and Emotion Recognition subscales) - change at 6 months | post-training (approximatively at month 6)
  The Theory of Mind and Affect Recognition subscales of NEPSY II are performance-based subtests aimed at evaluating social perception. They are administered to adolescents. Theory of Mind subscale-part A raw scores range from 0 to 17, Theory of Mind subscale-part b raw scores range from 0 to 8. Theory of Mind total subscale raw scores range from 0 to 25. Affect Recognition subscale raw scores range from 0 to 35. Raw scores are converted in scaled scores ranging from 1 to 19. Higher scores mean better outcomes.
A Developmental NEuroPSYchological Assessment-II (NEPSY-II) (Theory of Mind and Emotion Recognition subscales) - change at 12 months | post-training (approximatively at month 12)
  The Theory of Mind and Affect Recognition subscales of NEPSY II are performance-based subtests aimed at evaluating social perception. They are administered to adolescents. Theory of Mind subscale-part A raw scores range from 0 to 17, Theory of Mind subscale-part b raw scores range from 0 to 8. Theory of Mind total subscale raw scores range from 0 to 25. Affect Recognition subscale raw scores range from 0 to 35. Raw scores are converted in scaled scores ranging from 1 to 19. Higher scores mean better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute IRCCS E. Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No